CLINICAL TRIAL: NCT02698618
Title: PRotective Effect on the Coronary Microcirculation of Patients With DIabetes by Clopidogrel or Ticagrelor
Acronym: PREDICT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundacion Investigacion Interhospitalaria Cardiovascular (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Javier Escaned, Unit head, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-15-10793; 2015-003621-33 (EudraCT Number)
Record Dates: First submitted 2016-02-11; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; IMR; Microcirculation; Ticagrelor; CFR; FFR; Coronary microcirculation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Random Allocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental): A loading dose of Ticagrelor 180mg followed by a dose of 90mg b.i.d. (during 48 hours)
  Interventions: Procedure: Diagnostic; Drug: Randomization; Procedure: PCI
- Clopidogrel (Active Comparator): A loading dose of Clopidogrel 600mg followed by a daily dose (during at least 48 hours) of 75mg
  Interventions: Procedure: Diagnostic; Drug: Randomization; Procedure: PCI

INTERVENTIONS:
Procedure: Diagnostic — Pre-PCI and treatment:
  1. At hospital admission: all consecutive patients referred for coronary angiography in stable ischemic heart disease will undergo a complete physical examination, Electrocardiogram (ECG) and laboratory blood testing including cardiac troponin and kinase mioband. Subjects will be investigated to confirm or diagnose existing diabetic or pre-diabetic status.
  2. At the time of diagnostic catheterization After informed consent, diabetic or pre-diabetic patients with at least one stenosis with a Fractional Flow Reserve value (FFR) ≤ 0.80 fulfilling all the inclusion/exclusion criteria will be included in the trial.At the same time, a multimodal physiology assessment, including Coronary Flow Reserve (CFR) and Index of Microcirculatory Resistance (IMR) will be measured.
Drug: Randomization — Randomization: patients will be randomly assigned (with 1:1 ratio) to receive either Clopidogrel or Ticagrelor before their clinically-indicated Percutaneous Coronary Intervention (PCI). Either a loading dose of Ticagrelor 180mg followed by a dose of 90mg b.i.d. (during 48 hours) or a loading dose of Clopidogrel 600mg followed by a daily dose (during at least 48 hours) of 75mg will be administered according to their randomization. Additionally the groups will be balanced according to obesity prevalence [Body Mass Index (BMI) ≥30 kg/m2] with the implementation of a dedicated randomization list.
Procedure: PCI — 1. Pre-PCI: multimodal physiological evaluation: FFR, CFR, IMR will be repeated
  2. PCI: For all the patients undergoing PCI, the use of unfractioned heparin (UHF) will be allowed at the time of PCI; UFH be administered with a target on Activated Clotting Time (ACT) of 200-250 s. The PCI procedures will be performed by standard technique using only second generation Drug Eluting Stents (DES). In all cases, balloon pre-dilatation will be performed before stent implantation using a semi-compliant balloon with a diameter lower than a 75% of the distal reference diameter of the vessel to avoid confounders Post-dilation will be performed according to clinical practice although it will be not mandatory.
  3. Post-PCI: After stent implantation/s, multimodal physiological evaluation will be re-performed (FFR, CFR, IMR).

SUMMARY:
The purpose of this study is to determine whether Ticagrelor has a protective effect on microcirculation during percutaneous coronary interventions in patients with Diabetes mellitus type II or in a pre-diabetic status.

DETAILED DESCRIPTION:
Introduction:

Patients with Diabetes Mellitus (DM) Type 2 still consistently perform worse than their non-diabetic counterparts especially in the setting of Percutaneous Coronary Intervention (PCI). The abnormal coronary microcirculation along with the higher risk of distal embolization of particles released from the PCI target lesion constitutes the main cause of peri-procedural microcirculatory damage.

New antiplatelet agents, in particular Ticagrelor, might also play a protective role on microcirculation. Ticagrelor inhibits cellular uptake of adenosine, increasing the circulating levels of adenosine through the inhibition of its physiological clearance. Adenosine may protect the myocardium from both ischemic, and reperfusion injury via its potent vasodilatory effects and possibly by anti-inflammatory and antiplatelet properties.

Additionally previous research have identified a more profound effect of adenosine on microcirculatory resistance associated to obesity and diabetes and a higher myocardial protective effect of Ticagrelor during PCI might be expected in this high risk subgroup of patients.

The purpose of PRotective Effect on the Coronary Microcirculation of Patients With DIabetes by Clopidogrel or Ticagrelor (PREDICT) trial was designed to investigate the protective effect of Ticagrelor on microcirculation during PCI in stable diabetic patient

Rationale:

1. Coronary plaques at high risk for distal embolization during PCI, like the one with thin-cap fibroatheroma (TCFA), are more prevalent in patient with DM. Thus, this population is at high risk to develop myocardial injury and microcirculation impairment subsequent to PCI.
2. By blocking the Adenosine transporter (ENT) 1 nucleoside cell membrane transporter, Ticagrelor inhibits cellular uptake of adenosine, increasing the circulating levels of adenosine through the inhibition of its physiological clearance. Adenosine may protect the myocardium from both ischemic, and reperfusion injury via its potent vasodilatory effects and possibly by anti-inflammatory and antiplatelet properties. This translates into an adenosine-mediated vasodilatory effect of ticagrelor that takes place soon after loading dose.
3. Previous research from our group have identified a more profound effect of adenosine on microcirculatory resistance associated to obesity and diabetes and a higher myocardial protective effect of Ticagrelor during PCI might be expected in this high risk subgroup of patients. (enhanced microcirculatory response to raised adenosine levels).

Giving these premises in diabetics or pre-diabetics patients, Ticagrelor treatment pre-PCI might improve microcirculatory parameters (lower resistance) compared with clopidogrel (secondary hypothesis). Ticagrelor might be superior to clopidogrel in providing microcirculatory protection during PCI procedures in the same subgroup of patients (primary hypothesis).

ELIGIBILITY:
Inclusion Criteria:

* Subject with Diabetes Mellitus (DM) Type II
* Subject must be older than 18 years
* Written informed consent available
* Subject with stable ischemic heart disease referred for coronary angiography
* Subject is eligible for PCI, and PCI target(s) have FFR≤0.80

Exclusion Criteria:

* Prior myocardial infarction in the territory of the target vessel
* Akinesia or dyskinesia in subtended myocardial segments
* Severe impairment of left ventricular function (LVEF) <35%
* PCI target is a chronic total occlusion
* Target lesion has been treated previously (restenotic lesions)
* Target vessel is a saphenous vein graft or a surgical graft has been anastomosed to target vessel
* Thrombolisis in Myocardial Infarction (TIMI) flow ≤ 1 prior to guide wire crossing
* Subject is not eligible for treatment with DES
* Bleeding disorders or chronic anticoagulant treatment
* Left main stenosis > 50%
* Coronary surgery deemed more beneficial for the patient than PCI
* Intolerance or contraindications to anti-platelet drugs
* Contraindications for adenosine administration
* Platelet count <75000 or >700000/mm3
* Immunosuppressive therapy
* Pregnant or breast feeding patient
* History of intracranial haemorrhage
* Severe hepatic impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Delta IMR post-PCI | at least 48 hours after randomization, just after PCI and stenting.
  Absolute difference in the IMR value associated to PCI ["Delta IMR Post-PCI" = (IMR value post-PCI) minus (IMR value pre-PCI)]
Delta IMR pre-PCI | at least 48 hours after randomization, just before PCI and stenting.
  Absolute difference in the IMR value associated to PCI ["Delta IMR Pre-PCI" = (IMR value pre-PCI) minus (IMR value at baseline)]

SECONDARY OUTCOMES:
Myocardial necrosis associated to PCI damage | at least 72 hours, at the time of hospital discharge.
  Myocardial necrosis associated to PCI damage, assessed by cardiac markers (troponin rise > 5 times 99th percentile of upper reference limit or as elevation of CK-MB 3 times the upper limit of normal
IMR post-PCI | at least 48 hours after randomization, just after PCI and stenting.
  Absolute resistance value after PCI
Severe microcirculatory impairment | at least 48 hours after randomization, just after PCI and stenting.
  Incidence of severe microcirculatory impairment defined as Index of Microvascular Resistance > 29 after PCI

OTHER OUTCOMES:
Delta IMR post-PCI in subject with BMI = or > 30 | at least 48 hours after randomization, just after PCI and stenting.
  Absolute difference in the IMR value associated to PCI ["Delta IMR Post-PCI" = (IMR value post-PCI) minus (IMR value pre-PCI)] in subject with BMI = or > 30
Delta IMR pre-PCI in subject with BMI = or > 30 | at least 48 hours after randomization, just before PCI and stenting.
  Absolute difference in the IMR value associated to PCI ["Delta IMR Post-PCI" = (IMR value post-PCI) minus (IMR value pre-PCI)] in subject with BMI = or > 30
Myocardial necrosis associated to PCI damage in subject with BMI = or > 30 | at least 72 hours, at the time of hospital discharge.
  Myocardial necrosis associated to PCI damage, assessed by cardiac markers (troponin rise > 5 times 99th percentile of upper reference limit or as elevation of CK-MB 3 times the upper limit of normal in subject with BMI = or > 30
IMR post-PCI in subject with BMI = or > 30 | at least 48 hours after randomization, just after PCI and stenting.
  Absolute resistance value after PCI in subject with BMI = or > 30
Severe microcirculatory impairment in subject with BMI = or > 30 | at least 48 hours after randomization, just after PCI and stenting.
  Incidence of severe microcirculatory impairment defined as Index of Microvascular Resistance > 29 after PCI in subject with BMI = or > 30

CONTACTS AND LOCATIONS:
Overall Officials: Javier Escaned, MD, PhD, Principal Investigator — Hospital San Carlos, Madrid, Spain; Enrico Cerrato, MD, Principal Investigator — San Luigi Gonzaga University Hospital, Orbassano (Turin), Italy
Locations (3):
- Spain (3):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital San Carlos, Madrid, Madrid
  - Hospital Galdakao-Usansolo, Bilbao, Vizcaya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cerrato E, Quiros A, Echavarria-Pinto M, Mejia-Renteria H, Aldazabal A, Ryan N, Gonzalo N, Jimenez-Quevedo P, Nombela-Franco L, Salinas P, Nunez-Gil IJ, Rumoroso JR, Fernandez-Ortiz A, Macaya C, Escaned J. PRotective Effect on the coronary microcirculation of patients with DIabetes by Clopidogrel or Ticagrelor (PREDICT): study rationale and design. A randomized multicenter clinical trial using intracoronary multimodal physiology. Cardiovasc Diabetol. 2017 May 19;16(1):68. doi: 10.1186/s12933-017-0543-5. PMID 28526024